CLINICAL TRIAL: NCT07237360
Title: Impact in Pediatric Emergency Departments of a Systematic Individualized Interview Conducted by an Advanced Practice Nurse, on the Prevention of Safe Sleeping and Unexpected Infant Death, in a Population of Infants From 0 to 6 Months
Brief Title: Impact of Prevention of Safe Sleeping and Unexpected Infant Death
Acronym: MinUTE
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC25_0113
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Unexpected Infant Death; Prevention & Control; Safe Sleeping

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Emergencies babies
  Interventions: Other: Sleeping mode

INTERVENTIONS:
Other: Sleeping mode — Smoking habits, socio-professional category

SUMMARY:
The sudden unexpected infant death (SUID) is defined as "the sudden death of a child aged from 1 month to 1 year who had been healthy until then, whereas nothing in his known history or in the history of events could have allowed him to predict". In France, the French High Autority of Health (Haute Autorité de Santé (HAS)) has set the upper age limit at 2 years.

According to french statistics, between 250 and 350 babies die each year of unexpected infant death. It is the leading cause of infant mortality in developed countries, with all the devastating psychological, social and legal consequences for families. The national prevention campaigns for the "back to sleep" SUID carried out in the 1990s allowed a 75% decrease in the number of SUID. Yet, still at the moment, around 150 deaths could be avoided each year in France by respecting strict dorsal sleeping recommendations and a safe environment.

According to the SUID register of Nantes (France) of April 2024, 75% of deaths occur before the child's six months. The risk factors are mainly prematurity, exposure to tobacco (during and after pregnancy), and a sleeping mode not recommended by HAS. Indeed, on the day of death, 20% of babies were lying on their stomach or side, 30% shared their bed and 59% were lying in bedding at risk of containment or obstruction of the upper airway.

According to the database of National Association of Infant Death Unexpected Reference Centers since 2022, there has been a resurgence in the number of these deaths. This proves the urgency of prevention on this public health issue.

In parallel, we do not know why the number of SUID is not decreasing in correlation with the decrease in the birth rate in France. Moreover, it would be interesting to know the reasons why parents do not follow the recommendations of the HAS for their baby to sleep safely.

Thus, I wish to evaluate the impact of systematic prevention by the Advanced Practice Nurse with the parents of infants aged 0 to 6 months presenting to the Pediatric Emergency and know their barriers/levers to change.

My research question is therefore titled:

Why and how many infants under 6 months sleep in insecurity compared to lying babies according to the international recommendations ?

ELIGIBILITY:
Inclusion Criteria:

* All parents consulting the Pediatric Emergency Department of University Hospital of Angers for their baby aged 0 to 6 months

Exclusion Criteria:

* Any other person consulting for a baby aged 0 to 6 months who is not the parent of the baby: a grandparent, an uncle, an aunt, a childminder, the nursery manager, a friend of the parents, etc.
* Parent refusing the use of their data
* Parent and/or child under legal protection
* Parent who does not understand French

Ages: 0 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Parents of children from 0 to 6 months consulting at the Pediatric Emergency Department of University Hospital of Angers.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Increase in the number of babies lying well on their backs after the guided interview VS the number of babies lying well on their backs before the guided interview | During the interview of the family, about 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No